CLINICAL TRIAL: NCT02525146
Title: Birmingham Access to Care Study
Acronym: BA2C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Birmingham AIDS Outreach (Unknown); Johns Hopkins University (Other); AIDS United (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F130522004
Record Dates: First submitted 2015-08-01; First posted 2015-08-17 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: HIV Infection; HIV Care Loss to Followup
Keywords: HIV; Reengagement in HIV Care; ARTAS
MeSH Terms: conditions — HIV Infections | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients randomized to the intervention arm receive intensive social work case management based on the ARTAS (Antiretroviral Treatment and Access to Services) model. Patients may participate in 6-12 visits over a six-month period aimed at addressing barriers to re-engagement in HIV care. Participants complete a battery of research questions at Baseline, 6-months, and 12-months and HIV-1 viral load and CD4 count labwork at Baseline and at 12-months post enrollment.
  Interventions: Other: Modified ARTAS (Antiretroviral Treatment and Access to Services) intervention
- Usual Care (No Intervention): Patients randomized to the usual care arm are provide contact information for an HIV primary care clinic and for local AIDS service organizations. Patients are then encouraged to contact these organizations to re-establish care. Participants complete a battery of research questions at Baseline, 6-months, and 12-months and HIV-1 viral load and CD4 count labwork at Baseline and at 12-months post enrollment. Patients in the usual care arm are offered the intensive casework intervention after their 12-month followup is complete.

INTERVENTIONS:
Other: Modified ARTAS (Antiretroviral Treatment and Access to Services) intervention
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether a modified form of the ARTAS (Antiretroviral Treatment and Access to Services) intervention, adapted for HIV patients who have fallen out of care, can be successful in re-engaging patients in care and reducing HIV-1 viral load.

ELIGIBILITY:
Inclusion Criteria:

* HIV patient with at least one primary care appointment since 1/1/10 but currently lost to follow-up defined as 1) currently out of care for greater than 7 months or 2) does NOT have two or more completed clinic visits separated by three or more months in time during a 12-month observation period (HRSA-HAB measure of retention in care) or 3) has 2 or more "no shows" - scheduled visits for which the patient has not arrived or canceled - in the past 12 months.
* 19 years or older
* Be able and willing to provide informed consent
* Be willing to provide locator information
* Be willing to sign a HIPAA authorization form/medical record release form to facilitate medical record abstraction
* Report living in the vicinity
* Be able to communicate in English.

Exclusion Criteria:

* Not meeting one of the above inclusion criteria
* Have significant cognitive or developmental impairment to the extent that they are unable to provide informed consent
* Incarcerated at the time of potential enrollment
* Are terminated via site PI decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in HIV-1 Viral Load from Baseline to 12-month Followup | Baseline and 12-month Followup
  HIV-1 viral load is obtained via study-specific lab work done at Baseline and at the 12-month followup session.

SECONDARY OUTCOMES:
Re-Engagement in Care: Post-Enrollment Linkage Visit + Meeting HRSA-HAB Guidelines for Retention in Care | 12-month
  Using HIV primary care clinic attendance records, participants are assessed as to 1) whether or not an HIV Primary Care visit was completed post study enrollment and 2) following that visit, whether the participant made and kept appointments as necessary to meet HRSA-HAB guidelines constituting retention in HIV care. BOTH conditions must be present in order for participant to be considered "re-engaged" in care.

CONTACTS AND LOCATIONS:
Overall Officials: James L Raper, PhD, CRNP, JD, Principal Investigator — University of Alabama at Birmingham, 1917 HIV Clinic; Michael J Mugavero, MD, MHSc, Study Director — University of Alabama at Birmingham; David S Batey, PhD, MSW, LCSW, Study Director — University of Alabama at Birmingham